CLINICAL TRIAL: NCT01459094
Title: Single-Dose, Open-Label, Randomized, 2-Period Crossover Study to Assess the Effect of Food Coadministration on the Pharmacokinetics of a Fixed Dose Combination Tablet of Canagliflozin and Metformin Immediate Release in Healthy Subjects
Brief Title: Effect of Food on a Fixed Dose Combination Tablet of Canagliflozin and Metformin Immediate Release in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100652; 28431754DIA1037 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Oral bioavailability; Canagliflozin (JNJ-28431754); Metformin IR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence AB (Experimental)
  Interventions: Drug: A (CANA/MET IR FDC tablet - fasting state) / B (CANA/MET IR FDC tablet - fed state)
- Treatment Sequence BA (Experimental)
  Interventions: Drug: B (CANA/MET IR FDC tablet - fed state) / A (CANA/MET IR FDC tablet - fasting state)

INTERVENTIONS:
Drug: A (CANA/MET IR FDC tablet - fasting state) / B (CANA/MET IR FDC tablet - fed state) — Treatment A: Type = 1, unit = mg, number = 150/1000, form = tablet, route = oral use. One CANA/MET IR FDC tablet taken orally (by mouth) in a fasting state on Day 1 of Treatment Period 1 followed 10-14 days later by Treatment B: Type = 1, unit = mg, number = 150/1000, form = tablet, route = oral use. One CANA/MET IR FDC tablet taken orally in a fed state on Day 1 of Treatment Period 2.
  Arms: Treatment Sequence AB
Drug: B (CANA/MET IR FDC tablet - fed state) / A (CANA/MET IR FDC tablet - fasting state) — Treatment B: Type = 1, unit = mg, number = 150/1000, form = tablet, route = oral use. One CANA/MET IR FDC tablet taken orally in a fed state on Day 1 of Treatment Period 1 followed 10-14 days later by Treatment B: Type = 1, unit = mg, number = 150/1000, form = tablet, route = oral use. One CANA/MET IR FDC tablet taken orally in a fasting state on Day 1 of Treatment Period 2.
  Arms: Treatment Sequence BA

SUMMARY:
The purpose of this study is to see if the absorption and distribution of a fixed-dose Combination (FDC) tablet of canagliflozin and metformin IR is affected when taken with food by healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label (identity of study drug will be known to volunteers and study staff), single-center study to evaluate the oral bioavailability (ie, absorption and distribution within the body) and pharmacokinetics (blood levels) of a single dose of 1 fixed-dose combination (FDC) tablet of canagliflozin and metformin IR (abbreviated as 1 CANA/MET IR FDC tablet) when taken by healthy volunteers without food (in a fasting state) or with food (in a fed state). Healthy volunteers participating in the study will be randomly (by chance) assigned to receive Treatment A (1 CANA/MET IR FDC tablet taken by healthy volunteers in a fasting state) followed approximately 14 days later by Treatment B (1 CANA/MET IR FDC tablet taken by healthy volunteers in a fed state) or Treatment B followed approximately 14 days later by Treatment A.

ELIGIBILITY:
Inclusion Criteria: - Body mass index (BMI) between 18 and 30 kg/m² inclusive and a body weight of not less than 50 kg. Exclusion Criteria: - History of or current medical illness, abnormal values for hematology or clinical chemistry laboratory tests, or abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) deemed to be clinically significant by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Canagliflozin plasma concentrations | Up to 72 hours
Metformin plasma concentrations | Up to 24 hours

SECONDARY OUTCOMES:
Adverse events | Up to approximately 22 days
  The number and type of adverse events will be reported from Day 1 of treatment period 1 through 7-10 days after treatment period 2 including the 10-14 day washout period between treatment periods (total time is approximately 22 days).
Clinical Laboratory Tests | Up to approximately 22 days
  Clinically relevant changes from baseline occurring in laboratory safety parameters
Vital Signs | Up to approximately 22 days
  Changes from baseline in blood pressure and pulse

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC L.LC. Clinical Trial, Study Director — Janssen Research & Development, LLC

REFERENCES:
- [Derived] Murphy J, Wang SS, Stieltjes H, Wajs E, Devineni D. Effect of food on the pharmacokinetics of canagliflozin/metformin (150/1,000 mg) immediate-release fixed-dose combination tablet in healthy participants. Int J Clin Pharmacol Ther. 2015 Mar;53(3):256-64. doi: 10.5414/CP202233. PMID 25546166